CLINICAL TRIAL: NCT02124317
Title: Phase II Trial of Nab-paclitaxel Plus S-1 in First-line Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: Nab-paclitaxel Plus S-1 in Patients With Advanced Pancreatic Cancer
Acronym: NAPSPAC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dai, Guanghai, Professor and chief physician, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABXS001
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Advanced Pancreatic Cancer
Keywords: nanoparticle albumin-bound paclitaxel; S-1; advanced pancreatic cancer; objective response rate
MeSH Terms: interventions — Taxes; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- nanoparticle albumin-bound paclitaxel, S-1 (Experimental): nanoparticle albumin-bound paclitaxel is given at 120 mg/m2 intravenously on day 1 and 8, in combination with S-1 which is orally administered (40-60 mg according to the body surface, twice a day) on day 1-14 of each 21 day cycle. Number of cycle: 6 cycles.
  Interventions: Drug: nanoparticle albumin-bound paclitaxel; Drug: S-1

INTERVENTIONS:
Drug: nanoparticle albumin-bound paclitaxel — nanoparticle albumin-bound paclitaxel is given at 120 mg/m2 intravenously on day 1 and 8 of each 21 day cycle. Number of cycles: 6 cycles.
  Other Names: nab-paclitaxel; Abraxane; ABI-007
Drug: S-1 — S-1 is orally administered (40-60 mg according to the body surface, twice a day) on day 1-14 of each 21 day cycle. Number of cycles: 6 cycles.

SUMMARY:
The purpose of this study is to determine the efficacy and safety of nanoparticle albumin-bound paclitaxel (nab-paclitaxel) plus S-1 as first-line treatment in Chinese patients with advanced pancreatic ductal adenocarcinoma (PDA).

DETAILED DESCRIPTION:
Advanced PDA is a lethal disease with a approximately 6 months of median survival. Gemcitabine is always the only approved single agent. The recent results of the phase III trial MPACT (Metastatic Pancreatic Adenocarcinoma Clinical Trial) demonstrated an improvement in overall response rate (ORR), progression free survival (PFS) and overall survival (OS) for the combination of nab-paclitaxel plus gemcitabine compared to gemcitabine alone. Thus, the combination of nab-paclitaxel with gemcitabine became one of a standard treatment in metastatic PDA. S-1 is an oral fluoropyrimidine, and shown to be non-inferior to gemcitabine on OS for unresectable pancreatic cancer, and also demonstrated non-inferior, and even superior to gemcitabine as adjuvant chemotherapy. This single-arm study is to explore the efficacy and safety of nab-paclitaxel plus S-1 as first-line treatment in Chinese patients with local advanced or metastatic pancreatic ductal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed-consent form.
2. Age no less than 18 years.
3. Histologically confirmed locally advanced or metastatic pancreatic ductal adenocarcinoma, with RECIST measurable lesions.
4. Eastern Cooperative Oncology Group (ECOG) 0-1 with life expectation of no less than 12 weeks.
5. Patients must have received no previous chemotherapy or investigational therapy for the treatment of metastatic disease. Prior treatment with 5-fluorouracil or gemcitabine administered as a radiation sensitizer in the adjuvant setting is allowed, provided at least 6 months have elapsed since completion of the last dose and no lingering toxicities are present.
6. Adequate liver/bone marrow function.
7. Human Chorionic Gonadotropin (HCG) test negative for female with contraception measure until 3 months after study end.
8. Compliant, and can be followed up regularly.

Exclusion Criteria:

1. Pregnant or breast-feeding female, or not willing to take contraception measures during study.
2. Serious infection requiring antibiotics intervention during recruitment.
3. Allergic to study drug.
4. More than grade 1 neuropathy.
5. Uncontrolled brain metastasis or mental illness.
6. Congestive heart failure, uncontrolled cardiac arrhythmia, etc.
7. Other malignancy within 5 years.
8. Can't be followed up or obey protocol.
9. Ineligible by the discretion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Measure at every 6 weeks (every 2 cycles)
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST).

SECONDARY OUTCOMES:
Progression-free survival | up to 15 months
  Measure of time from study treatment to disease progression or death.
Overall survival | up to 2 years
  Measure of time from study treatment to patient's death or lost to follow-up.
Disease control rate | Measure every 6 weeks (every 2 cycles)
  The sum of rates of partial response, complete response and steady disease based on Response Evaluation Criteria In Solid Tumors (RECIST).
Safety and tolerability | up to 18 month
  Percentage of patients who experience adverse events during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Guanghai Dai, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Shi Y, Zhang S, Han Q, Li J, Yan H, Lv Y, Shi H, Liu R, Dai G. Nab-paclitaxel plus S-1 in advanced pancreatic adenocarcinoma (NPSPAC): a single arm, single center, phase II trial. Oncotarget. 2017 Sep 28;8(54):92401-92410. doi: 10.18632/oncotarget.21359. eCollection 2017 Nov 3. PMID 29190925